CLINICAL TRIAL: NCT00003008
Title: Pilot Study to Evaluate the Potential Interactions Between Paclitaxel and Protease Inhibitors in Patients With AIDS-Related Kaposi's Sarcoma
Brief Title: Paclitaxel in Treating Patients With AIDS-Related Kaposi's Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); AIDS Associated Malignancies Clinical Trials Consortium (Other)
Responsible Party: Group Chair, Eastern Cooperative Oncology Group
Purpose: Treatment
Other Study IDs: CDR0000065583; E1D95; AMC-014
Record Dates: First submitted 1999-11-01; First posted 2003-07-11 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Sarcoma
Keywords: AIDS-related Kaposi sarcoma; recurrent Kaposi sarcoma
MeSH Terms: conditions — Sarcoma; AIDS-related Kaposi sarcoma; Sarcoma, Kaposi | interventions — Indinavir; Nelfinavir; Paclitaxel; Ritonavir; Saquinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: indinavir sulfate
Drug: nelfinavir mesylate
Drug: paclitaxel
Drug: ritonavir
Drug: saquinavir mesylate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of paclitaxel in treating patients with AIDS-related Kaposi's sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether the body distribution and plasma clearance of paclitaxel is affected by protease inhibitors (e.g., indinavir, ritonavir, saquinavir mesylate, or nelfinavir mesylate).

OUTLINE: Patients are stratified according to protease inhibitor treatment (yes vs no), prior paclitaxel (yes vs no), and prior doxorubicin or daunorubicin (yes vs no).

Patients receive paclitaxel IV over 3 hours on day 1. Treatment continues every 2 weeks for at least 1 course in the absence of disease progression or unacceptable toxicity. Patients who previously received paclitaxel receive no more than 1 course during this study.

PROJECTED ACCRUAL: A total of 33 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Kaposi's sarcoma requiring chemotherapy and/or currently being treated with paclitaxel
* Serologic diagnosis of HIV infection documented by a positive ELISA and confirmed with a Western Blot or other federally approved HIV diagnostic test

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm ^3(with or without the use of colony-stimulating factors)
* Platelet count at least 50,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Neurologic:

* No greater than grade 2 peripheral neuropathy
* No neuropsychiatric history or altered mental status that would preclude study

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other prior or concurrent malignancy except curatively treated carcinoma in situ of the cervix or basal cell or squamous cell skin cancer
* No sensitivity to E. coli-derived proteins
* No active untreated infection
* No new infectious complications requiring a change in antibiotics within the past 2 weeks

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 1 week since prior radiotherapy
* No prior radiotherapy to marker lesions
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* At least 2 weeks since prior systemic treatment for Kaposi's sarcoma
* At least 2 weeks since prior nonapproved FDA investigational agents except available Investigational New Drugs that are antiretroviral agents
* Concurrent maintenance therapy for opportunistic infections allowed
* Concurrent commercially available antiretroviral therapy allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 1997-12-15 (Actual); Primary Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Hayden Von Roenn, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama, United States